CLINICAL TRIAL: NCT01813279
Title: Assessment of the Subcutaneous Reinjection of Human Autologous Adipose-derived Stromal Vascular Fraction (Celution® System) in the Hands of Patients Suffering From Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A01228-33; 2011-28 (Other: AP HM)
Record Dates: First submitted 2013-02-22; First posted 2013-03-18 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients (Experimental)
  Interventions: Other: the cell therapy

INTERVENTIONS:
Other: the cell therapy — the reinjection of autologous stromal vascular fraction of adipose tissue issue on the fingers of patients with scleroderma.

SUMMARY:
Systemic sclerosis is an autoimmune disease characterized by skin lesions and visceral responsible for significant morbidity. Microcirculatory disorders and tissue fibrosis are excessive severity of the disease. This condition can affect the hands with a major functional consequence severely impairing the quality of life of patients.

Adipose tissue is used in plastic surgery for over a century for the filling of depressions in the skin. In addition to the volume effect, a trophic effect on the surrounding tissue was noted. It is shown that the stromal vascular fraction is responsible for this regenerative effect.

In a previous study the investigators have demonstrated in a mouse model that the subcutaneous adipose tissue provides a trophic effect on SSc skin lesions by reducing the fibrosis of the dermis and providing a pro angiogenic.

Objectives and means:

This is a clinical study evaluating an innovative cell therapy procedure. The objective of this study was to evaluate the effects of injection of autologous stromal vascular fraction of adipose origin according to the system Celution ® (Cytori Therapeutics, Inc.., United Kingdom) in digital in patients with scleroderma cutaneous hands.

Eleven patients with scleroderma with the hands will be included in the study. Due to the nature of the orphan disease, a longitudinal study be conducted, where each patient will have own control.

The evaluation will be pre and post operative for a period of six months. This evaluation will be based on clinical criteria (trophic balance, functional) and laboratory (capillaroscopy, Doppler ultrasound of the arteries of the forearm, laser-Doppler tissue).

Project schedule and implementation phases:

The project will run over a period of twelve months. Patients will be followed for a period of six months. Analyzes clinical, paraclinical, and exploitation of results will be achieved over a period of six months.

Expected Results: This study will validate the functional and trophic effects of reinjection of autologous stromal vascular fraction of adipose tissue issue on the fingers of patients with scleroderma.

Conclusion: This innovative cell therapy could represent an alternative treatment for patients with scleroderma in check, intolerant or insufficiently relieved by medical treatment currently available in the scleroderma hand

ELIGIBILITY:
Inclusion Criteria:

* Men and women of more than 18 years old wishing a therapeutic alternative.
* Functional Disability of the hand authenticated by a functional index of the hand of Cochin upper to 20.

Exclusion Criteria:

* Persons participating simultaneously in another biomedical search(research)
* Minors
* Pregnant or breast-feeding Women
* Major Persons protected by the law (under guardianship or guardianship)
* Persons staying in a sanitary or social establishment
* Persons in emergency situation
* Private persons of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The improvement of the functional index of Cochin | 2 years

SECONDARY OUTCOMES:
Analog visual scale ( EVA ) | 24 MONTHS
Evaluation of the severity of the syndrome of Raynaud | 24 months
The test HAMIS | 24 months
The score of Rodnan modified in the hand | 24 months
-The test HAMIS | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: loic MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Granel B, Daumas A, Jouve E, Harle JR, Nguyen PS, Chabannon C, Colavolpe N, Reynier JC, Truillet R, Mallet S, Baiada A, Casanova D, Giraudo L, Arnaud L, Veran J, Sabatier F, Magalon G. Safety, tolerability and potential efficacy of injection of autologous adipose-derived stromal vascular fraction in the fingers of patients with systemic sclerosis: an open-label phase I trial. Ann Rheum Dis. 2015 Dec;74(12):2175-82. doi: 10.1136/annrheumdis-2014-205681. Epub 2014 Aug 11. PMID 25114060